CLINICAL TRIAL: NCT05104723
Title: A Phase 1/2 Open-label Study to Evaluate the Safety and Efficacy of Tofacitinib for Chronic Granulomatous Disease With Inflammatory Complications
Brief Title: Safety and Efficacy of Tofacitinib for Chronic Granulomatous Disease With Inflammatory Complications
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000064; 000064-I
Record Dates: First submitted 2021-11-02; First posted 2021-11-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-05-07

CONDITIONS: Chronic Granulomatous Disease; Inflammatory Gastrointestinal Disease; Inflammatory Skin Disease; Inflammatory Lung Disease
Keywords: Inflammatory Bowel Disease; Interferon (IFN)-induced gene expression; JAK Inhibitor; Ulcerative Colitis; Inflammatory skin/ lung disease
MeSH Terms: conditions — Granulomatous Disease, Chronic; Dermatitis; Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XELJANZ (tofacitinib) (Experimental): Tofacitinib is self-administered orally at 5 mg twice per day or 11 mg once per day for 3 months.
  Interventions: Drug: XELJANZ (tofacitinib)

INTERVENTIONS:
Drug: XELJANZ (tofacitinib) — The XELJANZ 5-mg tablets or 11-mg XR tablets will taken orally twice daily or once daily, respectively, in this study.

SUMMARY:
Background:

Chronic granulomatous disease (CGD) is a disease of the immune system, which is how the body fights germs. People with CGD get infections easily and have other health problems. Some medicines to treat CGD have a lot of side effects and do not always work. Researchers want to see if a new drug can help.

Objective:

To see if tofacitinib is safe to use for treating chronic CGD.

Eligibility:

Adults aged 18 and older with CGD who have not had success with other treatments and who are enrolled on NIH study # 93-I-0119.

Design:

Participants will be screened with the following:

Physical exam

Medical history

Blood, urine, and stool tests

Pregnancy test, if needed

An upper gastrointestinal endoscopy and/or colonoscopy, if needed for their symptoms. Tissue samples will be collected.

Skin assessment, if needed

Participants will repeat some screening tests at visits.

Participants will complete questionnaires about their general health and how CGD affects their daily life. Photographs will be taken of their skin, if needed. They will have lung function tests, if needed. They will have a computed tomography (CT) scan of the chest, abdomen, and pelvis, if needed. A CT scan uses X-rays to create pictures of the inside of the body.

Participants will gradually reduce the amount of some CGD medicines they take. Then they will take tofacitinib as a pill twice a day or once a day for 3 months. They will keep a drug diary. They will have monthly study visits. They will have a follow-up visit about 1 month after their last study drug visit.

Participation will last for about 6 months.

DETAILED DESCRIPTION:
Study Description:

This is a phase 1/2 open-label trial to study the safety and to explore the biological efficacy of tofacitinib in patients with confirmed and symptomatic inflammatory complications (gastrointestinal [GI], skin, lung) related to chronic granulomatous disease (CGD). After a 3-month regimen, participants inflammatory complications will be objectively assessed.

Primary Objective:

To assess the safety of tofacitinib during the study period in patients with CGD.

Secondary Objectives:

1. To assess the overall clinical response for the specific inflammatory manifestations.
2. To assess the biological effect of tofacitinib on interferon (IFN)-induced gene expression in CGD.

Primary Endpoints:

1. Rate of infection.
2. Rate of treatment-related toxicities.
3. Rate of adverse events (AEs).
4. Incidence of serious bacterial, mycobacterial, fungal, or viral infections defined as infections that require medical assessment or hospitalization.

Secondary Endpoints:

CGD-related inflammatory bowel disease (IBD):

1. Change in modified Harvey-Bradshaw Index (HBI).
2. Change in histopathological endoscopy.

Inflammatory lung disease:

1. Change in forced expiratory volume (FEV1).
2. Change in diffusing capacity for carbon monoxide (DLCO).
3. Change in computed tomography (CT) radiography.
4. Change in 6-minute walk.

Skin disease:

1. Change in presence of skin flares or ulcerations by objective photography evaluation.

Gene expression:

1.Change in IFN gene module enrichment score derived from whole blood RNA expression data.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Aged >=18 years.
2. Enrolled on NIH study 93-I-0119.
3. Has a documented diagnosis of one or more of the following and is not controlled under current therapy (per investigator assessment):

   1. Endoscopically diagnosed mild-to-severe CGD-related IBD.
   2. Radiographic or PFT changes (DLCO<60%, FEV1<70%) consistent with CGD-related inflammatory lung disease.
   3. Any inflammatory skin disease related to CGD (eg, hidradenitis suppurativa or granulomatous skin disease).
4. Able to provide informed consent.
5. Participants who can become pregnant or who can impregnate their partner must agree to use at least one highly effective method of contraception when engaging in sexual activities that can result in pregnancy, starting at the first dose of tofacitinib until 2 days after the last dose. Highly effective methods include a barrier (eg, condom, diaphragm, cervical cap), intrauterine device, or hormonal contraception.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known allergy or hypersensitivity to any component of the tofacitinib formulation.
2. Known allergy or hypersensitivity to any component of the acyclovir or valacyclovir formulation.
3. Active or latent tuberculosis.
4. Infection with hepatitis B or C, or HIV.
5. Active EBV infection.
6. History of GI perforation.
7. History of malignancy (except for nonmelanoma skin cancer).
8. Concomitant use of acetylsalicylic acid and/or NSAIDs that cannot be safely discontinued.
9. History of connective tissue disease.
10. End-stage renal disease or chronic kidney disease, defined as estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m^2.
11. Evidence of other invasive or systemic fungal, bacterial, or viral infections requiring therapy.
12. Pregnant.
13. Breastfeeding.
14. Current use of inhaled tobacco products, vaping product, inhaled cannabis, or other illicit inhaled drugs.
15. Current use of strong CYP3A4 inducer and unable to discontinue at least 14 days before beginning of tofacitinib regimen.
16. Concomitant medical condition that could interfere with study drug evaluation or that is a contraindication to the proposed investigational treatment based upon known agent safety profile or toxicities.
17. Any of the following laboratory abnormalities:

    1. Alkaline phosphatase and either ALT or AST >2.5 times the upper limit of normal (ULN).
    2. Serum creatinine level >5 mg/dL.
    3. Absolute neutrophil count (ANC) <1000 cells/microL.
    4. Lymphocyte count <500 cells/microL.
18. History of unprovoked deep vein thrombosis, pulmonary embolism, or other thrombotic events.
19. History of heart failure.
20. Current immobilization, ie, bed-bound and unable to ambulate.
21. Exposure to any investigational agent within the last 4 weeks.
22. Any other finding that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant s ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment-related toxicities. | Day 1 through Day 120
  To assess the safety of tofacitinib during the study period in patients with CGD.
Rate of infection. | Day 1 through Day 120
  To assess the safety of tofacitinib during the study period in patients with CGD.
Rate of AEs | Day 1 through Day 120
  To assess the safety of tofacitinib during the study period in patients with CGD.
Incidence of serious bacterial, mycobacterial, fungal, or viral infections defined as infections that require medical assessment or hospitalization. | Day 1 through Day 120
  To assess the safety of tofacitinib during the study period in patients with CGD.

SECONDARY OUTCOMES:
CGD-related IBD: 1.Change in modified HBI. 2.Change in histopathological endoscopy. | Day 90
  To assess the overall clinical response for the specific inflammatory manifestations.
Skin disease: 1.Change in presence of skin flares or ulcerations by objective photography evaluation. | Day 90
  To assess the overall clinical response for the specific inflammatory manifestations.
Inflammatory lung disease: 1. Change in FEV1. 2. Change in DLCO. 3.Change in CT radiography. 4. Change in 6-minute walk. | Day 90
  To assess the overall clinical response for the specific inflammatory manifestations.
Gene expression: 1.Change in IFN gene module enrichment score derived from whole blood RNA expression data. | Day 90
  To assess the biological effect of tofacitinib on IFN-induced gene expression in CGD.

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panes J, Sandborn WJ, Schreiber S, Sands BE, Vermeire S, D'Haens G, Panaccione R, Higgins PDR, Colombel JF, Feagan BG, Chan G, Moscariello M, Wang W, Niezychowski W, Marren A, Healey P, Maller E. Tofacitinib for induction and maintenance therapy of Crohn's disease: results of two phase IIb randomised placebo-controlled trials. Gut. 2017 Jun;66(6):1049-1059. doi: 10.1136/gutjnl-2016-312735. Epub 2017 Feb 16. PMID 28209624
- [Background] Henrickson SE, Jongco AM, Thomsen KF, Garabedian EK, Thomsen IP. Noninfectious Manifestations and Complications of Chronic Granulomatous Disease. J Pediatric Infect Dis Soc. 2018 May 9;7(suppl_1):S18-S24. doi: 10.1093/jpids/piy014. PMID 29746679
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000064-I.html